CLINICAL TRIAL: NCT00199589
Title: Treatment of Spastic Equinovarus Foot After Stroke. Efficacy: Association Between Ankle Foot Orthosis and Botulinum Toxin A (BTA) Injection
Brief Title: Treatment of Spastic Equinovarus Foot After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Allergan (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I01014
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: Spastic Equinovarus
Keywords: Spastic equinovarus; Botox; Ankle foot orthosis
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Botulinic toxin (Botox) — Patients may benefit, depending on the draw, in addition to their orthosis, intramuscular injections of botulinum toxin.These injections are among 6 in the muscles posterior (rear) of the leg paralyzed with tracking electromyographic to ensure the accuracy of the injection.

SUMMARY:
This study evaluates treatment for spastic foot after stroke using ankle foot orthosis with or without selective injection of BTA (Botox).

DETAILED DESCRIPTION:
This prospective, multicentric open trial evaluates the efficacy of a combined treatment for spastic foot after stroke using ankle foot orthosis with or without selective injection of BTA (Botox) into the tibialis anterior and/or posterior and/or the long toe flexor, and/or medial and lateral gastrocnemius, and/or soleus muscles [300 BTA U per injection (Botox - Allergan), diluted with saline to a concentration of 5U/0,1 mL, with electromyography guided injection]. The patients are followed for one year after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stroke patient with equinovarus foot due to severe lower limb extensor spasticity with impaired foot contact during walking
* Ability to walk for at least 10 meters with or without aid
* Stroke interval < 12 months
* Age > 18 years old
* Weight > 30 kg and < 100 kg
* Written informed consent

Exclusion Criteria:

* Stroke interval > 12 months
* Age < 18 years old
* Pregnancy
* Neuromuscular disease
* Previous treatment with BTA
* Fixed contractures impairing mobility
* Mini-Mental Status Examination < 25
* Aminosides treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2002-10; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Plantar contact during walking

SECONDARY OUTCOMES:
Gait velocity
Barthel index
MIF
Autosatisfaction by EVA
Asworth scale
Ankle range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Salle, MD, Principal Investigator — University Hospital, Limoges
Locations (2):
- France (2):
  - Département de Médecine Physique et de Réadaptation, Bordeaux
  - Département de Médecine Physique et de Réadaptation, CHU Limoges, Limoges